CLINICAL TRIAL: NCT06421441
Title: The Effect of Self-Management Skills Training Given to Nursing Students According to Peer Education Module on Problematic Internet Use and Academic Procrastination Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cennet Ciriş Yıldız, Dr. Faculty Member, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1919B012203792
Record Dates: First submitted 2023-01-30; First posted 2024-05-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Problem Behavior; Problematic Internet Use; Academic Procrastination Behavior
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: Group 1: Experimental group (Education group) Goup 2: Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Experimental group (Education group)
  Interventions: Other: Self Management Skills Training
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Self Management Skills Training — Nursing students will be given self-management skills training for a total of 12 hours, two days a week, two hours a day (60 min. + 60 min.) for three weeks.
  Arms: Experimental

SUMMARY:
The aim of the study is to evaluate the effect of self-management skills training given with the peer education module on the problematic internet use and academic procrastination behavior of nursing students. .

DETAILED DESCRIPTION:
A total of 12 hours of self-management skills training will be given to the peer groups, two days a week for three weeks, two lesson hours a day (60 min. + 60 min.).The effect of self-management skills training on problematic internet use and academic procrastination behavior of nursing students will be evaluated.

ELIGIBILITY:
Research Inclusion Criteria;

* Being 18 years or older,
* Volunteering to participate in the study,
* Using the internet for an average of 2 hours or more per day,
* Not having any communication problems,
* To continue self-management skills training.

Criteria for Exclusion from the Research;

* Having any communication barrier,
* Not continuing self-management skills training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Problematic Internet Use Scale | Before training, immediately in the first and third months after training
  It was developed in order to reveal the healthy and unhealthy usage levels of the Internet. The total score varies between 27 and 135. This scale aims to reveal healthy and unhealthy internet usage levels. In this context, high scores that can be obtained from the scale should be considered as a sign that individuals' internet use has become unhealthy, the internet has a negative impact on their lives, and may create a tendency towards a pathology such as addiction.
Academic Procrastination Scale | Before training, immediately in the first and third months after training.
  It was developed to determine students' academic procrastination behaviors. The highest score that can be obtained from the scale is 95 and the lowest score is 19. A high score from the scale indicates that students are academic procrastinators.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın Üniversity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided